CLINICAL TRIAL: NCT06551597
Title: The Effect of Extremely Low-Frequency Magnetic Field on Physical Fitness and Inflammatory Markers in Post-Stroke Patients
Brief Title: The Effect of Extremely Low-Frequency Magnetic Field on Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, dr n. o zdr. Trzmiel Tomasz, Assistant professor, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Magneto1
Record Dates: First submitted 2024-08-07; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: extremely low - frequency magnetic fields therapy; stroke; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MT1 - The group receiving magnetotherapy to the head in addition to standard therapy (Experimental)
  Interventions: Procedure: Extremely low frequency electromagnetic fields stimulation
- MT2 - The group receiving magnetotherapy to the pelvis in addition to standard therapy (Active Comparator)
  Interventions: Procedure: Extremely low frequency electromagnetic fields stimulation
- Control group - The group receiving only standard therapy (No Intervention)

INTERVENTIONS:
Procedure: Extremely low frequency electromagnetic fields stimulation — * In Group MT1, patients will undergo 10 sessions (over 10 consecutive days excluding weekends) of low-frequency magnetotherapy (exposure site - head, 40 Hz, 5 mT) as addition to standard neurological rehabilitation.
  * In Group MT2, patients will undergo 10 sessions (over 10 consecutive days excluding weekends) of low-frequency magnetotherapy (exposure site - pelvis, 40 Hz, 5 mT) as addition to standard neurological rehabilitation.
  * The control group participants will receive only neurological rehabilitation.
  Arms: MT1 - The group receiving magnetotherapy to the head in addition to standard therapy; MT2 - The group receiving magnetotherapy to the pelvis in addition to standard therapy

SUMMARY:
A stroke can cause neurological deficits resulting in decreased motor, sensory, and cognitive function, as well as a decline in psychosocial functioning. Early rehabilitation following a stroke incident is of great importance, and interventions should aim for an overall improvement in patient functioning and achieving the highest possible level of independence. In recent years, there has been an emphasis on the need to regulate the inflammation that occurs after a stroke, as it may influence the improvement or deterioration of the patient's condition. Initial studies have also indicated the potential for influencing post-stroke inflammation through physical therapy procedures. In studies on the impact of magnetotherapy on inflammatory processes in post-stroke patients, magnetotherapy is usually applied to the pelvic girdle or the head area. However, the effectiveness of these two application methods has not yet been compared. In this study, investigators aim to compare the effects of magnetotherapy applied to different body areas as a complement to neurological rehabilitation. The study aims to assess the impact of magnetotherapy as a complement to neurological rehabilitation on physical fitness and inflammatory markers in post-stroke patients, to evaluate the effect of magnetotherapy as a supplement to neurological rehabilitation on physical fitness and oxidative stress markers in post-stroke patients, and to assess the differences between the effects of magnetotherapy applied to the pelvic area versus magnetotherapy applied to the head area.

The participants will be divided into three groups: one will serve as the control group, while the other two will receive magnetotherapy to the head or the pelvis, respectively, as an addition to standard neurological therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Ischemic stroke within a maximum of two weeks prior to admission to the ward

Exclusion Criteria:

* Severe functional impairment (FIM score < 37)
* History of previous strokes
* Other neurological diseases or other conditions that could significantly impair the patient's functioning
* Contraindications to magnetotherapy
* Inability to establish logical verbal communication with the patient
* Lack of informed consent to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure | The study will be conducted on the day of admission, after the series of treatments (approximately on the 14th day of stay), and at the day of discharge (approximately on the 35th day of stay)
  The Functional Independence Measure (FIM) is a standardized tool used to assess a person's level of independence in performing daily activities, including self-care, mobility, and communication, with the results expressed in points.The total score for the FIM instrument will range between 18 and 126. he higher the score, the more independent the patient is.
Barthel Scale | The study will be conducted on the day of admission, after the series of treatments (approximately on the 14th day of stay), and at the day of discharge (approximately on the 35th day of stay)
  The Barthel Scale is a standardized tool used to measure a person's ability to perform basic activities of daily living independently, such as feeding, bathing, dressing, and mobility, with the results expressed in points. The score can range from 0 to 100, with 100 indicating the highest level of patient independence.
Tinetti Scale | The study will be conducted on the day of admission, after the series of treatments (approximately on the 14th day of stay), and at the day of discharge (approximately on the 35th day of stay)
  The Tinetti Scale is a standardized assessment tool used to evaluate a person's balance and gait, helping to determine their risk of falling, with the results expressed in points.
  The Tinetti Scale is scored from 0 to 28 points, with lower scores indicating a higher risk of falls.
Berg Balance Scale | The study will be conducted on the day of admission, after the series of treatments (approximately on the 14th day of stay), and at the day of discharge (approximately on the 35th day of stay)
  The Berg Balance Scale is a standardized tool used to assess a person's balance through various tasks, helping to evaluate their risk of falling, with the results expressed in points. Berg balance scale scores range from 0 to 56. The lower is the score, the higher is the risk of loosing balance and fall.
Short Physical Performance Battery | The study will be conducted on the day of admission, after the series of treatments (approximately on the 14th day of stay), and at the day of discharge (approximately on the 35th day of stay)
  The Short Physical Performance Battery (SPPB) is a standardized tool used to assess lower extremity function through a series of tasks, including balance, walking speed, and chair stands, with the results expressed in points. The scores range from 0 (worst performance) to 12 (best performance).

SECONDARY OUTCOMES:
C-reactive protein | The study will be conducted on the day of admission, after the series of treatments (approximately on the 14th day of stay), and at the day of discharge (approximately on the 35th day of stay)
  C-reactive protein (CRP) is a blood test used to measure the level of inflammation in the body, which can indicate the presence and severity of infection or other inflammatory conditions, with the results expressed in milligrams per liter (mg/L)
Procalcitonin blood levels ng/ml | The study will be conducted on the day of admission, after the series of treatments (approximately on the 14th day of stay), and at the day of discharge (approximately on the 35th day of stay)
  Procalcitonin is a blood test used to assess the level of procalcitonin, a biomarker that helps indicate the presence and severity of bacterial infections, particularly sepsis. It is also an important marker of the inflammatory process and oxidative stress in stroke patients, with the results expressed in nanograms per milliliter (ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Hojan, Assoc Prof, Study Director — Poznan University of Medical Sciences
Locations (1):
- Neurorehabilitation Ward, Greater Poland Provincial Hospital, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No